CLINICAL TRIAL: NCT03167411
Title: A Phase 1, Open-label, Randomized, Two-period, Two-treatment, Crossover Study to Evaluate the Effect of Exenatide on the Pharmacokinetics and Pharmacodynamics of Bexagliflozin in Healthy Subjects
Brief Title: Bexagliflozin Drug/Drug Interaction Study With Exenatide Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-458
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-03

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — bexagliflozin; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bexagliflozin alone (Experimental)
  Interventions: Drug: Bexagliflozin
- Bexagliflozin with exenatide injection (Active Comparator)
  Interventions: Drug: Bexagliflozin; Drug: Exenatide Injection

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin tablets, 20 mg
Drug: Exenatide Injection — Byetta® (Exenatide), 10 ug, bid, subcutaneous injection
  Other Names: Byetta®
  Arms: Bexagliflozin with exenatide injection

SUMMARY:
The purpose of this study is to examine the drug-drug interaction when given the study drug, bexagliflozin, with one of the most commonly prescribed glucagon-like peptide 1 receptor agonist (GLP-1 RA) exenatide. The study will also evaluate how safe the study drug is and how well the study drug is tolerated when administered with exenatide injection.

DETAILED DESCRIPTION:
This was a phase 1, single center, open-label, 2 × 2 crossover study designed to assess the effects of exenatide injection on the PK and PD of orally administered bexagliflozin tablets. Healthy subjects were randomly assigned to one of two groups with 10 subjects per group. Each group received both the treatments, alternately, in a crossover fashion with the two treatment periods separated by a 7-day washout period.

In Treatment Period 1, subjects were admitted to the clinic on day 0, the day before dosing, and stayed in the clinic until 48 h post-dose. After an overnight fast of at least 10 h, subjects in Group 1 received a single oral dose of bexagliflozin tablets, 20 mg, alone 30 min before breakfast, and subjects in Group 2 received a subcutaneous (SC) injection of exenatide at 10 µg twice a day (bid) with an initial dose 30 min prior to a single oral dose of bexagliflozin tablets, 20 mg, and 1 hr before breakfast, followed by the second dose of exenatide alone 1 hr prior to the evening meal.

In Treatment Period 2, subjects were admitted to the clinic on day 7, the day before dosing, and stayed in the clinic until 48 hr post-dose. After an overnight fast of at least 10 h, subjects in Group 1 received a SC injection exenatide at 10 µg bid with an initial dose 30 min prior to a single oral dose of bexagliflozin tablets, 20 mg, and 1 hr before breakfast and followed by the second dose of exenatide alone 1 hr prior to the evening meal. Subjects in Group 2 received a single oral dose of bexagliflozin tablets, 20 mg, alone 30 minutes before breakfast.

Blood samples for bexagliflozin plasma concentration were collected during each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 hr post-dose. Pre-dose urine samples were collected from -12 to 0 hr for baseline measurement of PD parameters. Post-dose urine samples were collected in four batches: 0 to 12 hr, 12 to 24 hr, 24 to 36 hr, and 36 to 48 hr.

Clinical laboratory tests and safety monitoring were conducted during both treatment periods for each group.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects who were between the ages of 18 and 65 years, inclusive, in good health based on medical history, physical examination, electrocardiogram and routine laboratory tests.
2. Subjects with body-mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2, inclusive.
3. Subjects who were non-smokers for at least 3 months prior to screening.
4. Subjects with adequate venous access at multiple sites in both arms.
5. Subjects who were willing and able to be confined to the clinical research facility as required by the protocol.
6. Subjects who had the ability to comprehend and who were willing to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

1. Subjects who were determined by the investigator or sub-investigator to be unsuitable for participation in the study based on medical conditions or factors that would have influenced adherence to study activities.
2. Subjects with a clinically significant history of allergy to drugs or latex.
3. Subjects with a history of hypoglycemia.
4. Subjects with a history of alcohol or drug dependence in the last 12 months.
5. Subjects who donated 400 mL of whole blood within 56 days, 200 mL of whole blood within one month, or donated blood components within 14 days of screening.
6. Subjects who used prescription or over-the-counter (OTC) drugs within 14 days prior to the first dose.
7. Subjects who used vitamin preparations or supplements (including St. John's Wort and ginseng) within 14 days prior to the first dose .
8. Subjects who were not willing to refrain from smoking, alcohol, grapefruit, grapefruit juice or related products, caffeine consumption (including chocolate), and strenuous exercise within 72 h prior to Day 1 and through the end of the PK study.
9. Male subjects who did not agree to refrain from donating sperm and use appropriate birth control methods including condoms with spermicide, female partner's use of diaphragm with spermicide, or stable oral, implanted, or injected contraceptive hormones, or with an intrauterine device, or female partner is surgically sterile (i.e. have undergone partial or full hysterectomy, or bilateral oophorectomy) or postmenopausal (absence of menses greater than 12 months and age >45 years), for a period of 30 days after discharge from the clinic.
10. Female subjects of childbearing potential who were not willing to use an adequate method of contraception including bilateral tubal ligation, intrauterine device, diaphragm with spermicide and male partner's use of male condom with spermicide, and to not become pregnant for the duration of the study. Female subjects who were surgically sterile (partial or full hysterectomy, or bilateral oophorectomy) or postmenopausal (absence of menses greater than 12 months and age >45 years) were eligible if they tested negative on the pregnancy test.
11. Subjects who had been treated with an investigational drug within 30 days or 7 half-lives of the investigational drug, whichever is longer, prior to the first dose of study drug in this trial.
12. Subjects who had previously received exenatide, or any other GLP-1 RAs within three months from the screening or subjects who had had any GLP-1 RA and suffered an adverse reaction due to the medication.
13. Subjects who had previously received bexagliflozin, or any other SGLT2 inhibitors within 3 months from the screening.
14. Subjects whose screening ECG demonstrates any one of the following: heart rate >100 bpm, QRS >120 msec, QTc >470 msec (corrected by Fridericia's formula), PR >220 msec (a subject with PR >220 msec was generally to be excluded but exceptions may have been allowed at the discretion of the investigator), or any clinically significant arrhythmia.
15. Subjects whose sitting blood pressure was above 140/90 mmHg at screening. If the sitting blood pressure at screening was above 140/90 mmHg, one repeat measurement was allowed and the subject may have been randomized if the blood pressure was 140/90 +/-5 mm Hg at the discretion of the Investigator.
16. Subjects who had a positive result of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, urinary drug or urinary cotinine test.
17. Subjects with human immunodeficiency virus (HIV) infection.
18. Subjects who had had a febrile illness within 5 days prior to the first dose of study medication.
19. Subjects vaccinated within 30 days (with the exception of the flu vaccine) prior to the first dose of investigational drug.
20. Subjects with a history of acute or chronic pancreatitis or gall stones.
21. Positive urine glucose at screening.
22. Subjects with estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2 or a history of kidney transplant.
23. Subjects with digestion problems, including gastroesophageal reflux disease, irritable bowel syndrome, gastroparesis, and any other disorder deemed by the investigator to be clinically significant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, M.D., Study Chair — Massachusetts General Hospital
Locations (1):
- Clinical Research Site, Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 healthy subjects were randomly assigned to one of the two groups (1 or 2) and will receive both treatments alternately, in a crossover fashion (two-period, two-treatment crossover design), with the two treatment groups separated by a 7-day washout period.
Groups:
- Bexagliflozin, Then Bexagliflozin With Exenatide: After an overnight fast, subjects received a single oral dose of bexagliflozin tablets, 20 mg alone 30 min before breakfast. After a washout period of 7 days, the subjects then received a subcutaneous injection of exenatide 10 µg at 30 min prior to a single oral dose of bexagliflozin, and 1 hr before breakfast and followed by the second dose of exenatide alone 1 hr prior to the evening meal.
- Bexagliflozin With Exenatide, Then Bexagliflozin Alone: Subjects received a subcutaneous injection of exenatide at 10 µg twice a day (bid) with an initial dose 30 min prior to a single oral dose of bexagliflozin tablets, 20 mg, and 1 hr before breakfast, followed by the second dose of exenatide alone 1 hr prior to the evening meal. After a washout period of 7 days, the subjects then received a single oral dose of bexagliflozin tablets, 20 mg alone 30 min before breakfast.
Period: Overall Study
Arm/Group | Bexagliflozin, Then Bexagliflozin With Exenatide | Bexagliflozin With Exenatide, Then Bexagliflozin Alone
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bexagliflozin With Exenatide, Then Bexagliflozin: Subjects received a subcutaneous injection of exenatide at 10 µg twice a day (bid) with an initial dose 30 min prior to a single oral dose of bexagliflozin tablets, 20 mg, and 1 hr before breakfast, followed by the second dose of exenatide alone 1 hr prior to the evening meal. After a washout period of 7 days, the subjects then received a single oral dose of bexagliflozin tablets, 20 mg alone 30 min before breakfast.
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin, Then Bexagliflozin With Exenatide | Bexagliflozin With Exenatide, Then Bexagliflozin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (9.03) | 43.1 (14.79) | 39.1 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 6 | 7
  White | 6 | 4 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 77.6 (10.48) | 80.7 (17.29) | 79.1 (14.01)
Height [Mean (Standard Deviation); unit: cm] | 173.1 (9.66) | 170.8 (10.94) | 172.0 (10.11)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (3.45) | 27.3 (3.14) | 26.6 (3.29)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 109.1 (11.98) | 106.3 (8.11) | 107.7 (10.06)

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Plasma Concentration)
Description: Whole venous blood samples of 3 mL was collected from peripheral vein at each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose of bexagliflozin. A non-compartmental pharmacokinetic analysis was used to calculate the PK parameters. Cmax was obtained directly from experimental observations.
Time Frame: Up to 48 hrs
Population: Number of subjects in the PK population with data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Bexagliflozin: Bexagliflozin: Bexagliflozin tablets, 20 mg, oral, one dose
- Bexagliflozin With Exenatide: Bexagliflozin: Bexagliflozin tablets, 20 mg, oral, one dose
  Exenatide: Byetta® (Exenatide), 10 µg, subcutaneous injection, twice a day (bid), two doses
Arm/Group | Bexagliflozin | Bexagliflozin With Exenatide
Number analyzed (Participants) | 19 | 17
ng/mL | 95.9 (33.6) | 121.6 (33.1)
Statistical Analysis 1: Comparison: Bexagliflozin vs Bexagliflozin With Exenatide; Test type: Equivalence — The ratio of the least squares (LS) geometric means of Cmax when bexagliflozin is dosed in combination with exenatide versus when dosed alone, with 80-125% defined as the lack of interaction boundaries. 90% confidence intervals was constructed; Point Estimate (%) = 125.27, 90% CI 2-sided [104.45 to 150.24] — Estimated ratio (%) of exponentiated mean difference of log-transformed PK parameter from ANOVA (linear mixed-effects model), with treatment, period, and sequence as fixed effects, and subject as a random effect

2. Primary Outcome: Tmax (Time of Maximum Observed Plasma Concentration)
Description: Whole venous blood samples of 3 mL was collected from peripheral vein at each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose of bexagliflozin. A non-compartmental pharmacokinetic analysis was used to calculate the PK parameters. Tmax was obtained directly from experimental observations.
Time Frame: Up to 48 hrs
Population: Number of subjects in the PK population with data
Measure: Median (Full Range); unit: hours
Arm/Group | Bexagliflozin | Bexagliflozin With Exenatide
Number analyzed (Participants) | 19 | 17
hours | 2.00 [1 to 5] | 5.00 [2 to 10]

3. Primary Outcome: T1/2 (Apparent Terminal Elimination Half-life)
Description: Whole venous blood samples of 3 mL was collected from peripheral vein at each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose of bexagliflozin. A non-compartmental pharmacokinetic analysis was used to calculate the PK parameters. T1/2 was calculated as the natural log of 2 divided by the terminal phase rate constant.
Time Frame: Up to 48 hrs
Population: Number of subjects in the PK population with data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Bexagliflozin | Bexagliflozin With Exenatide
Number analyzed (Participants) | 16 | 16
hours | 12.1 (45.3) | 8.8 (31.5)

4. Primary Outcome: AUC0-inf (Area Under the Plasma Concentration-time Curve From Time 0 to Infinity)
Description: Whole venous blood samples of 3 mL was collected from peripheral vein at each period at pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36 and 48 h post-dose of bexagliflozin. A non-compartmental pharmacokinetic analysis was used to calculate the PK parameters. AUC0-inf was calculated using the linear trapezoidal rule, using actual elapsed time values. If the actual time of sample collection was not available, the nominal time was used for the purpose of parameter estimation.
Time Frame: Up to 48 hrs
Population: Number of subjects in the PK population with data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Bexagliflozin | Bexagliflozin With Exenatide
Number analyzed (Participants) | 16 | 16
hr*ng/mL | 776.0 (27.5) | 1085.3 (29.5)
Statistical Analysis 1: Comparison: Bexagliflozin vs Bexagliflozin With Exenatide; Test type: Equivalence — The ratio of the least squares (LS) geometric means of AUC0-inf when bexagliflozin is dosed in combination with exenatide versus when dosed alone, with 80-125% defined as the lack of interaction boundaries. 90% confidence intervals was constructed; Point Estimate (%) = 137.56, 90% CI 2-sided [122.28 to 154.75] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Urinary Glucose Excretion (UGE)
Description: Post-dose urine was collected without preservative in four batches: 0 to 12 h, 12 to 24 h, 24 to 36 h, and 36 to 48 h collections. After collection, the total volume of each batch and collection time was recorded. UGE, including UGE(t1-t2) and total 0-24 h and 0-48 h UGE were calculated. UGE(t1-t2) was derived from urine volume (Vt1-t2) multiplied by glucose concentration divided by 100.
Time Frame: 0-48 hours
Population: Number of subjects in the PD population with data in the specific category
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Bexagliflozin | Bexagliflozin With Exenatide
Number analyzed (Participants) | 19 | 17
g
  Pre-dose (-12 to 0 hours): number analyzed (Participants) | 18 | 16
  Pre-dose (-12 to 0 hours) | 0.07 (0.140) | 0.05 (0.100)
  0 - 12 hours | 38.32 (8.705) | 26.38 (8.347)
  12 - 24 hours: number analyzed (Participants) | 19 | 16
  12 - 24 hours | 26.89 (7.833) | 28.95 (6.812)
  24 - 36 hours | 21.93 (6.934) | 22.16 (6.845)
  36 - 48 hours | 9.56 (6.283) | 9.21 (6.499)
  0 - 24 hours: number analyzed (Participants) | 19 | 16
  0 - 24 hours | 65.21 (15.035) | 55.65 (12.123)
  0 - 48 hours: number analyzed (Participants) | 19 | 16
  0 - 48 hours | 96.70 (25.080) | 88.11 (20.525)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Day 0 to Day 10.
Arm/Group | Bexagliflozin | Bexagliflozin With Exenatide
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 4/20 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexagliflozin (N=20) | Bexagliflozin With Exenatide (N=20)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (7)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT03167411/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03167411/SAP_001.pdf